CLINICAL TRIAL: NCT02753517
Title: Predictive Value of Hepato Biliary Scintigraphy to Assess the Risk of Postoperative Liver Failure Hepatectomies Stretches of 4 or More Segments on Non-cirrhotic Liver
Brief Title: Hepato Biliary Scintigraphy to Assess the Risk of Postoperative Liver Failure Hepatectomies
Acronym: SCINTIVOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This premature termination was decided by the Sponsor due to the fact that the Cholediam required for the study had been unavailable for 2 years, with no visibility on its future availability.
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2014_02; 2014-A01685-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Insufficiency
Keywords: hepatobiliary scintigraphy; extended hepatectomy; volumetry
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extended hepatectomy (Other): Hepatic Scintigraphy
  Interventions: Device: Hepatobiliary scintigraphy

INTERVENTIONS:
Device: Hepatobiliary scintigraphy — hepatobiliary scintigraphy with functional assessment of the future remnant liver before an extended hepatectomy of 4 or more segments

SUMMARY:
Extended hepatectomies of 4 or more segments are complicated by high rates of morbidity and mortality, mainly related to hepatic liver failure. Nowadays, preoperative assessment of the future remnant liver is just performed through its volumetric measurement by computed tomography. Nevertheless, this volumetric assessment does not reflect the hepatocellular function of the future remnant liver that can be disturbed in case of vascular and/or biliary obstruction, chemotherapy-induced liver injuries or steatosis in overweight patients. Literature data (albeit originating from a single centre in Europe) have suggested that (99m)Tc-mebrofenin hepatobiliary scintigraphy could be useful in evaluating the function of the future remnant liver. The aim of this prospective multicentric study is to determine the predictive value of hepatobiliary scintigraphy in assessing the risk of postoperative liver failure of extended hepatectomies of 4 or more segments in noncirrhotic liver.

DETAILED DESCRIPTION:
The main aim of the study is to determine the predictive value of (99m)Tc-mebrofenin hepatobiliary scintigraphy in assessing the postoperative risk of liver failure within 3 months of extended hepatectomy of 4 or more segments in noncirrhotic liver. The main endpoint is the three-months postoperative liver failure, defined as an increased International Normalized Ratio (INR) and concomitant hyperbilirubinemia (according to the normal limits of the local laboratory) on or after postoperative day 5 according to the international classification of the ISGLS (International Study Group of Liver Surgery) and classified according to its severity in grade A (no change of the patient's clinical management), grade B (deviation from the regular course but without invasive therapy) and grade C (invasive treatment)

Secondary objectives are:

To determine the predictive value of (99m)Tc-mebrofenin hepatobiliary scintigraphy in assessing the risk of postoperative morbi-mortality (according to Clavien-Dindo classification) within 3 months of extended hepatectomy of 4 or more segments in noncirrhotic liver, and the duration of intensive care unit stay and of hospitalization.

* To assess the correlation between the results of the hepatobiliary scintigraphy and the presence of parenchymal abnormalities such as steatosis, fibrosis or chemotherapy-induced injuries (sinusoidal obstruction syndrome, steatohepatitis) at the histological analysis of the non tumoral liver parenchyma.
* To assess the sensitivity of hepatobiliary scintigraphy in jaundiced patients who had a preoperative biliary endoscopic or radiologic drainage, considering the existing competition between mebrofenin and bilirubin on hepatic receptors.
* To analyse the inter-centre reproducibility of the hepatobiliary scintigraphy (Central review by the principal investigator of 25 scintigraphy examinations per centre)

ELIGIBILITY:
Inclusion Criteria:

* Noncirrhotic liver
* Benign or malignant liver tumor
* Anatomic hepatic resection ≥ 4 segments
* Aged ≥18
* ASA Score ≤3
* Signed informed consent
* Presence of contraception in non-menopausal women

Exclusion Criteria:

* Cirrhosis
* Absence of preoperative biliary drainage in case of preoperative jaundice
* Patient refusal
* Absence of affiliation to Social Security
* Body weight above 230kg
* Known allergy to Hida derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Hepatic insufficiency | at 3 months
  ISGLS criteria : a definition and grading by the International Study Group of Liver Surgery (ISGLS)of the Posthepatectomy liver failure:

SECONDARY OUTCOMES:
Postoperative morbi-mortality | at 3 months
  Clavien-Dindo classification
Duration of intensive care unit stay and of hospitalization | 3 months
  Duration of hospitalization
Histological analysis of the non tumoral liver parenchyma | at 3 months
  correlation of liver parenchymal abnormalities with the results of scintigraphy
Inter-centre reproducibility of the hepatobiliary scintigraphy | at 3 months
  Central review by the principal investigator of 25 scintigraphy examinations per centre

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Truant, MD, Principal Investigator — University Hospital, Lille
Locations (12):
- France (12):
  - Hôpital Nord, CHU, Amiens
  - CHU, Bordeaux
  - Hopital Estaing - Chu63 - Clermont Ferrand, Clermont-Ferrand
  - CHU, Grenoble
  - CHRU, Hôpital Claude Huriez, Lille
  - Centre Leon Berard - Lyon 08, Lyon
  - Hopital Croix-Rousse - Hcl - Lyon 04, Lyon
  - CHU, Marseille
  - Chru Nancy - Hopitaux de Brabois, Nancy
  - AP-HPHôpital Beaujon,, Paris
  - CHU, Rouen
  - CHU, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bennink RJ, Tulchinsky M, de Graaf W, Kadry Z, van Gulik TM. Liver function testing with nuclear medicine techniques is coming of age. Semin Nucl Med. 2012 Mar;42(2):124-37. doi: 10.1053/j.semnuclmed.2011.10.003. PMID 22293167
- [Result] de Graaf W, Heger M, Spruijt O, Maas A, de Bruin K, Hoekstra R, Bennink RJ, van Gulik TM. Quantitative assessment of liver function after ischemia-reperfusion injury and partial hepatectomy in rats. J Surg Res. 2012 Jan;172(1):85-94. doi: 10.1016/j.jss.2010.06.038. Epub 2010 Jul 21. PMID 20869070
- [Result] de Graaf W, Bennink RJ, Vetelainen R, van Gulik TM. Nuclear imaging techniques for the assessment of hepatic function in liver surgery and transplantation. J Nucl Med. 2010 May;51(5):742-52. doi: 10.2967/jnumed.109.069435. Epub 2010 Apr 15. PMID 20395336
- [Result] de Graaf W, Hausler S, Heger M, van Ginhoven TM, van Cappellen G, Bennink RJ, Kullak-Ublick GA, Hesselmann R, van Gulik TM, Stieger B. Transporters involved in the hepatic uptake of (99m)Tc-mebrofenin and indocyanine green. J Hepatol. 2011 Apr;54(4):738-45. doi: 10.1016/j.jhep.2010.07.047. Epub 2010 Oct 1. PMID 21163547
- [Result] de Graaf W, van Lienden KP, van den Esschert JW, Bennink RJ, van Gulik TM. Increase in future remnant liver function after preoperative portal vein embolization. Br J Surg. 2011 Jun;98(6):825-34. doi: 10.1002/bjs.7456. Epub 2011 Apr 11. PMID 21484773